CLINICAL TRIAL: NCT03822026
Title: Effects of Moderate Hyperventilation on Cerebral Hemodynamics, Oxygenation and Metabolism in Patients With Severe Traumatic Brain Injury
Brief Title: Hyperventilation in Patients With Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEK-ZH 2012-0542 (1)
Record Dates: First submitted 2019-01-22; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Head Injury Trauma; Hyperventilation
Keywords: intracranial pressure; cerebral metabolism; cerebral oxygenation
MeSH Terms: conditions — Hyperventilation

STUDY DESIGN:
Intervention Model Description: several parameters are collected at different time points: at baseline conditions, during moderate hyperventilation, and after return to baseline
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with severe TBI (Other): Patients with severe TBI enrolled in the study undergo an hyperventilation test, in which the alveolar ventilation is increased by a stepwise increase in tidal volumes and respiratory rate until a reduction of etCO2 of 0.7 kPa is achieved.
  Interventions: Other: Hyperventilation test

INTERVENTIONS:
Other: Hyperventilation test — Increase of the alveolar ventilation by a stepwise increase in tidal volumes and respiratory rate until a reduction of end-tidal CO2 of 0.7 kPa is achieved

SUMMARY:
Elevated intracranial pressure is a dangerous and potentially fatal complication after traumatic brain injury. Hyperventilation is a medical intervention to reduce elevated intracranial pressure by inducing cerebral vasoconstriction, which might be associated to cerebral ischemia and hypoxia.

The main hypothesis is that a moderate degree of hyperventilation is sufficient to reduce the intracranial pressure without inducing cerebral ischemia.

DETAILED DESCRIPTION:
In patients with severe traumatic brain injury (TBI), and with intracranial pressure-monitoring, brain tissue oxygen tension and/or microdialysis probes hyperventilation-tests are performed in the acute phase after trauma. Data are collected and TCCD measurements are performed at baseline, at the beginning of moderate hyperventilation, after prolonged moderate hyperventilation (for 50 minutes) and after return to baseline.

The present study aims to quantify potential adverse effects of moderate short-term hyperventilation during the acute phase of the severe TBI on cerebral hemodynamics, oxygenation, and metabolism.

ELIGIBILITY:
Inclusion Criteria:

* nonpenetrating traumatic brain injury
* Glasgow coma scale <9 at presentation
* Intracranial pressure monitoring
* brain tissue oxygen tension monitoring and/or microdialysis monitoring
* invasive mechanical ventilation with FIO2 <60% and PEEP <15 mbar

Exclusion Criteria:

* decompressive craniectomy
* pregnancy
* pre-existing neurological disease
* previous traumatic brain injury
* acute cardiovascular disease
* severe respiratory failure
* acute on chronic liver disease
* sepsis
* failure to obtain satisfactory bilateral TCCD signals
* persisting hypovolemia or hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-05-20 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

PRIMARY OUTCOMES:
intracranial pressure | 10, 20, 50, 60 minutes after begin of the hyperventilation test
  Change of intracranial pressure during moderate hyperventilation

SECONDARY OUTCOMES:
cerebral flow velocity in the middle cerebral artery | 20, 50, 60 minutes after begin of the hyperventilation test
  Change of cerebral flow velocity during moderate hyperventilation
brain tissue oxygenation (PbrO2) | 10, 20, 50, 60 minutes after begin of the hyperventilation test
  no changes
cerebral Lactate/ Pyruvate ratio | 1 hour before initiation of the hyperventilation test, and 1 and 2 hours after begin of the hyperventilation test
  no changes

CONTACTS AND LOCATIONS:
Overall Officials: Peter Steiger, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Klinzing S, Stretti F, Pagnamenta A, Bechir M, Brandi G. Transcranial color-coded duplex sonography assessment of cerebrovascular reactivity to carbon dioxide: an interventional study. BMC Neurol. 2021 Aug 7;21(1):305. doi: 10.1186/s12883-021-02310-9. PMID 34364365
- [Derived] Brandi G, Stocchetti N, Pagnamenta A, Stretti F, Steiger P, Klinzing S. Cerebral metabolism is not affected by moderate hyperventilation in patients with traumatic brain injury. Crit Care. 2019 Feb 13;23(1):45. doi: 10.1186/s13054-018-2304-6. PMID 30760295